CLINICAL TRIAL: NCT00614679
Title: A Novel Catheter Lock Solution for Treatment of Tunneled Hemodialysis Catheter-Associated Bacteremia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Saima Aslam, Associate Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-17624
Record Dates: First submitted 2008-02-11; First posted 2008-02-13 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: End-Stage Renal Disease; Hemodialysis Catheter-associated Infection
Keywords: biofilm; catheter lock solution; catheter salvage
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Tigecycline; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): single arm trial of experimental catheter lock solution
  Interventions: Drug: catheter lock solution consisting of N-acetylcystein, tigecycline and heparin

INTERVENTIONS:
Drug: catheter lock solution consisting of N-acetylcystein, tigecycline and heparin — N-acetylcystein 80 mg/ml, tigecycline 1 mg/ml, and heparin 2000 units/ml. This will be a 5 ml catheter lock solution

SUMMARY:
The primary objective is to investigate the ability of systemic intravenous antibiotic plus antibiotic/anti-biofilm (i.e. N-acetylcysteine) lock catheter technique in eradicating uncomplicated catheter associated bacteremia and salvaging the infected vascular catheter. Secondary objectives include duration to clearance of bacteremia, future recurrence of bacteremia, need for catheter removal and death.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who have an indwelling hemodialysis catheter for 10 or more days and evidence of a catheter associated bloodstream infection as evidenced by 1)quantitative blood cultures obtained through the lumen of the catheter yield concentrations of bacterial colonies that are 5 or more fold higher than peripheral blood cultures, or 2)blood cultures obtained through the lumen of the catheter becomes positive 2 or more hours earlier than peripheral blood cultures.

Exclusion Criteria:

* Patients will be excluded if 1) they are unable or unwilling to provide informed consent, 2) have evidence of a complicated bacteremia such as endocarditis, septic thrombophlebitis, septic emboli, osetoemylitis, deep seated abscesses etc 3)evidence of an exit site infection around the catheter such as a pus pocket, drainage or erythema. 4) patient is allergic to NAC or the proposed antibiotic (if patient is allergic to minocycline, tigecycline will not be used). 5) patient is pregnant or will become pregnant.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-10; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Treatment success within 90 days | 90 days

SECONDARY OUTCOMES:
catheter salvage | 90 days

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Ben Taub General Hospital, Houston, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - The Methodist Hospital, Houston, Texas

REFERENCES:
- [Derived] Aslam S, Trautner BW, Ramanathan V, Darouiche RO. Pilot trial of N-acetylcysteine and tigecycline as a catheter-lock solution for treatment of hemodialysis catheter-associated bacteremia. Infect Control Hosp Epidemiol. 2008 Sep;29(9):894-7. doi: 10.1086/590192. PMID 18643743